CLINICAL TRIAL: NCT04953923
Title: A Randomized, Double-blinded, Double-dummy, Placebo-controlled Thorough QTC Study With Single Oral Doses of Cedazuridine in Healthy Subjects
Brief Title: Thorough QT Assessment of Cedazuridine in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astex Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: E7727-02
Record Dates: First submitted 2021-06-30; First posted 2021-07-08 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — cedazuridine; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Treatment A (Experimental): Cedazuridine at a therapeutic dose
  Interventions: Drug: Cedazuridine
- Treatment B (Experimental): Cedazuridine at a supratherapeutic dose
  Interventions: Drug: Cedazuridine
- Treatment C (Placebo Comparator): Placebo control
  Interventions: Drug: Placebo
- Treatment D (Active Comparator): Moxifloxacin positive control
  Interventions: Drug: Moxifloxacin

INTERVENTIONS:
Drug: Cedazuridine — Tablet for oral administration
  Arms: Treatment A; Treatment B
Drug: Placebo — Capsule for oral administration
  Arms: Treatment C
Drug: Moxifloxacin — Tablet for oral administration
  Arms: Treatment D

SUMMARY:
This study is designed to evaluate the effect of therapeutic and supratherapeutic oral doses of cedazuridine on cardiac repolarization, as detected by QTc in healthy subjects, in accordance with regulatory guidelines. Moxifloxacin will be used to validate the study. Study duration per participant is approximately 20 days.

ELIGIBILITY:
Inclusion Criteria:

* Male or female who is not of childbearing potential
* Body mass index of 18.0 to 32.0 kg/m^2, inclusive

Exclusion Criteria:

* QTcF >450 msec at screening
* Clinically relevant abnormalities in conduction parameters; or if PR interval > 200 msec, QRS duration > 110 msec, or bradycardia or tachycardia (HR <45 bpm or >100 bpm)
* History or presence of hypokalemia, hypomagnesemia, or hypocalcemia
* Risk factors for Torsades de Pointes (TdP) (eg, congenital deafness, heart failure, cardiomyopathy, concomitant medications known to cause QTc prolongation) within a washout of at least 30 days
* Family history of Long QT Syndrome or family history of TdP
* Sick sinus syndrome, atrioventricular block (any degree)
* Myocardial infarction, pulmonary congestion, cardiac arrhythmia, prolonged QT interval, or conduction abnormalities
* Repeated or frequent syncope or vasovagal episodes
* Resuscitated arrest possibly due to TdP; hypertension, angina, or severe peripheral arterial circulatory disorders
* Use of concomitant medications that prolong the QT/QTc interval

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2021-11-16 (Actual)

PRIMARY OUTCOMES:
Change from baseline in QTcF | Baseline and Day 20
  Change from baseline in QTcF following single therapeutic and supratherapeutic doses of cedazuridine

SECONDARY OUTCOMES:
Change from baseline in QTcF | Baseline and Day 20
  Change from baseline in QTcF following cedazuridine-epimer and moxifloxacin administration
Safety: Participants with adverse events | Up to Day 20
  Number of participants with adverse events following single therapeutic and supratherapeutic doses of cedazuridine
Change from baseline in heart rate | Baseline and Day 20
  Change from baseline in heart rate following single therapeutic and supratherapeutic doses of cedazuridine
Change from baseline in PR interval of the electrocardiogram (ECG) | Baseline and Day 20
  Change from baseline in PR interval of the ECG following single therapeutic and supratherapeutic doses of cedazuridine
Change from baseline in QRS interval of the electrocardiogram (ECG) | Baseline and Day 20
  Change from baseline in QRS interval of the ECG following single therapeutic and supratherapeutic doses of cedazuridine
Change from baseline in T-wave morphology | Baseline to Day 20
  Change from baseline in treatment-emergent T-wave morphology following single therapeutic and supratherapeutic doses of cedazuridine
Pharmacokinetic parameter: Cmax | Up to Day 20
  Cmax is the maximum observed plasma concentration of cedazuridine, cedazuridine-epimer, and moxifloxacin
Pharmacokinetic parameter: Tmax | Up to Day 20
  Tmax is the time to maximum observed plasma concentration of cedazuridine, cedazuridine-epimer, and moxifloxacin
Pharmacokinetic parameter: AUClast | Up to Day 20
  Area under the curve (AUC) from time 0 to time of last measurable concentration of cedazuridine, cedazuridine-epimer, and moxifloxacin

CONTACTS AND LOCATIONS:
Locations (1):
- PRA Health Sciences, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No